CLINICAL TRIAL: NCT03501277
Title: A Randomized, Open-Label, Single-Dose, 4-Period Crossover Study to Determine the Bioequivalence of Alogliptin (25 mg) and Pioglitazone (15 and 30 mg) When Administered as Individual Tablets and as Fixed-Dose Combination Tablets to Healthy Russian Subjects
Brief Title: A Study to Determine the Bioequivalence of Alogliptin and Pioglitazone When Administered as Individual Tablets and as Fixed-Dose Combination (FDC)-SYR-322-4833 BL Tablets to Healthy Russian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Alogliptin-1002; U1111-1196-9223 (Other: WHO)
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sequence I: ABCD (Experimental): SYR-322-4833 BL (alogliptin 25 [milligram] mg and pioglitazone 15 mg) FDC tablet, orally, once, on Day 1 of Period 1 (Regimen A), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 15 mg tablet, orally, once, on Day 1 of Period 2 (Regimen B), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 30 mg) FDC tablet, orally, once, on Day 1 of Period 3 (Regimen C), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 30 mg tablet, orally, once, on Day 1 of Period 4 (Regimen D).
  Interventions: Drug: Alogliptin; Drug: Pioglitazone; Drug: SYR-322-4833 BL
- Sequence II: BCDA (Experimental): Alogliptin 25 mg tablet and pioglitazone 15 mg tablet, orally, once, on Day 1 of Period 1 (Regimen B), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 30 mg) FDC tablet, orally, once, on Day 1 of Period 2 (Regimen C), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 30 mg tablet, orally, once, on Day 1 of Period 3 (Regimen D), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 15 mg) FDC tablet, orally, once, on Day 1 of Period 4 (Regimen A).
  Interventions: Drug: Alogliptin; Drug: Pioglitazone; Drug: SYR-322-4833 BL
- Sequence III: CDAB (Experimental): SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 30 mg) FDC tablet, orally, once, on Day 1 of Period 1 (Regimen C), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 30 mg tablet, orally, once, on Day 1 of Period 2 (Regimen D), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 15 mg) FDC tablet, orally, once, on Day 1 of Period 3 (Regimen A), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 15 mg tablet, orally, once, on Day 1 of Period 4 (Regimen B).
  Interventions: Drug: Alogliptin; Drug: Pioglitazone; Drug: SYR-322-4833 BL
- Sequence IV: DABC (Experimental): Alogliptin 25 mg tablet and pioglitazone 30 mg tablet, orally, once, on Day 1 of Period 1 (Regimen D), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 15 mg) FDC tablet, orally, once, on Day 1 of Period 2 (Regimen A), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 15 mg tablet, orally, once, on Day 1 of Period 3 (Regimen B), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 30 mg) FDC tablet, orally, once, on Day 1 of Period 4 (Regimen C).
  Interventions: Drug: Alogliptin; Drug: Pioglitazone; Drug: SYR-322-4833 BL

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets.
Drug: Pioglitazone — Pioglitazone tablets.
Drug: SYR-322-4833 BL — SYR-322-4833 BL FDC tablets.
  Other Names: Incresync

SUMMARY:
The purpose of this study is to assess the relative bioavailability and bioequivalence of 2 strengths of the FDC tablet product SYR-322-4833 BL compared to the individual alogliptin and pioglitazone tablets in healthy Russian participants.

DETAILED DESCRIPTION:
The drug being tested in this study are called Incresync (SYR-322-4833 BL), alogliptin, and pioglitazone. This study will assess the bioequivalence, pharmacokinetics (PK), and safety of alogliptin and pioglitazone administered as individual tablets and as the FDC tablet product in healthy volunteers.

The study will enroll approximately 72 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the 4 treatment sequences to receive one of the following treatments:

* Regimen A: SYR-322-4833 BL (25 mg + 15 mg)
* Regimen B: Alogliptin 25 mg + pioglitazone 15 mg
* Regimen C: SYR-322-4833 BL (25 mg + 30 mg)
* Regimen D: Alogliptin 25 mg + pioglitazone 30 mg

All participants will be asked to take single dose of study medication on Day 1 of each intervention period.

This single center trial will be conducted in Russia. The overall time to participate in this study is 66 days. Participants will make multiple visits to the clinic, and will be contacted by telephone 14 days after their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female.
2. Has an estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 90 milliliter per minute (mL/min).
3. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 18.5 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.

Exclusion Criteria:

1. Has participated in a clinical study within 3 months prior to Check-in (Day-1).
2. Has a fasting blood glucose level lower than 3.88 millimole per liter (mmol/L).
3. Has received alogliptin or pioglitazone in a previous clinical study or as a therapeutic agent within 90 days prior to Check-in (Day-1).
4. Experienced acute infectious diseases within 4 weeks prior to Screening.
5. Has a positive urine drug result for super potent substances and drugs of abuse (defined as any illicit drug use) or positive alcohol breath test at Screening or Check-in (Day -1).
6. Consumes over 10 drinks weekly (1 drink is equivalent to 0.5 liters of beer, 200 milliliter (mL) of dry wine or 50 mL of ardent spirits) or has a history of alcoholism, drug and/or substance abuse.
7. Has a non-standard diet (example, vegetarian or vegan) or lifestyle (including night time work, extreme physical activity such as weights lifting), which may interfere with the trial.
8. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
9. Has poor peripheral venous access.
10. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1 of Period 1.
11. Has consumed caffeine or xanthine-containing food or drinks within 72 hours prior to Check-in (Day -1).
12. Has dehydration due to vomiting, diarrhea, or any other reason within 24 hours prior to study start.
13. Has drug intolerance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Non-governmental healthcare Institution Road Clinical Hospital at the station Yaroslavl JSC Russian Railways, Yaroslavl, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Russia from 26 May 2018 to 11 July 2018.
Pre-assignment Details: Healthy participants were enrolled in 1 of the 4 treatment sequences to receive: SYR-322-4833 BL (25 milligram [mg] + 15 mg) (Regimen A), alogliptin 25 mg + pioglitazone 15 mg (Regimen B), SYR-322-4833 (25 mg + 30 mg) (Regimen C), and alogliptin 25 mg + pioglitazone 30 mg (Regimen D).
Groups:
- Sequence I: ABCD: SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 15 mg) fixed dose combination (FDC) tablet, orally, once, on Day 1 of Period 1 (Regimen A), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 15 mg tablet, orally, once, on Day 1 of Period 2 (Regimen B), followed by a 7-day washout period, followed by SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 30 mg) FDC tablet, orally, once, on Day 1 of Period 3 (Regimen C), followed by a 7-day washout period, followed by alogliptin 25 mg tablet and pioglitazone 30 mg tablet, orally, once, on Day 1 of Period 4 (Regimen D).
Period: Intervention Period 1 (4 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 18 | 18
Safety Analysis Set | 18 | 18 | 17 | 17
Completed | 18 | 18 | 17 | 17
Not Completed | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout Period 1 (7 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 17 | 17
Completed | 18 | 18 | 17 | 17
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 2 (4 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 17 | 17
Completed | 18 | 18 | 17 | 16
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout Period 2 (7 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 17 | 16
Completed | 18 | 18 | 17 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 3 (4 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 17 | 16
Completed | 18 | 18 | 17 | 15
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout Period 3 (7 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 17 | 15
Completed | 18 | 18 | 17 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 4 (4 Days)
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC
Started | 18 | 18 | 17 | 15
Completed | 18 | 18 | 17 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence I: ABCD | Sequence II: BCDA | Sequence III: CDAB | Sequence IV: DABC | Total
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (7.95) | 23.9 (4.60) | 29.4 (8.46) | 27.5 (6.36) | 27.4 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 9 | 33
  Male | 9 | 11 | 9 | 8 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 17 | 17 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 18 | 18 | 17 | 17 | 70
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 18 | 18 | 17 | 17 | 70
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 68.77 (12.527) | 69.86 (12.409) | 75.06 (14.643) | 71.22 (15.894) | 71.17 (13.806)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.21 (3.411) | 24.06 (2.959) | 24.78 (3.575) | 24.89 (3.628) | 24.48 (3.342)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.3 (8.56) | 169.9 (8.02) | 173.6 (10.22) | 168.4 (9.44) | 170.0 (9.14)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Alogliptin and Pioglitazone
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all participants in the safety set who had sufficient plasma concentration data to facilitate the derivation of at least 1 PK parameter.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Groups:
- Regimen A: SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 15 mg) FDC tablet, orally, once, on Day 1 of Period 1, 2, 3 or 4.
- Regimen B: Alogliptin 25 mg tablet and pioglitazone 15 mg tablet, orally, once, on Day 1 of Period 1, 2, 3 or 4.
- Regimen C: SYR-322-4833 BL (alogliptin 25 mg and pioglitazone 30 mg) FDC tablet, orally, once, on Day 1 of Period 1, 2, 3 or 4.
- Regimen D: Alogliptin 25 mg tablet and pioglitazone 30 mg tablet, orally, once, on Day 1 of Period 1, 2, 3 or 4.
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 70 | 69 | 68 | 70
nanogram per milliliter (ng/ml)
  Alogliptin | 165.3 (42.87) | 154.9 (44.71) | 162.3 (51.19) | 157.4 (44.24)
  Pioglitazone | 678.3 (267.58) | 706.5 (254.12) | 1052.1 (478.13) | 1141.5 (509.78)
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; Test type: Equivalence — Alogliptin: For each analyte, an analysis of variance (ANOVA) was performed on natural logarithm transformed Cmax with factors for sequence, the participant nested within sequence, period, and regimen. For the relative bioavailability (BA) determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90 percent (%) confidence interval (CI) for the ratio of Cmax for Regimen A (test) versus Regimen B (reference); p = 0.014, ANOVA; Least Square Mean (LSM) difference = 1.0706, 90% CI 2-sided [1.0230 to 1.1204]
Statistical Analysis 2: Comparison: Regimen C vs Regimen D; Test type: Equivalence — Alogliptin: For each analyte, ANOVA was performed on natural logarithm transformed Cmax with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of Cmax for Regimen C (test) versus Regimen D (reference); p = 0.326, ANOVA; LSM difference = 1.0276, 90% CI 2-sided [0.9817 to 1.0757]
Statistical Analysis 3: Comparison: Regimen A vs Regimen B; Test type: Equivalence — Pioglitazone: For each analyte, ANOVA was performed on natural logarithm transformed Cmax with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of Cmax for Regimen A (test) versus Regimen B (reference); p = 0.405, ANOVA; LSM diiference = 0.9594, 90% CI 2-sided [0.8837 to 1.0415]
Statistical Analysis 4: Comparison: Regimen C vs Regimen D; Test type: Equivalence — Pioglitazone: For each analyte, ANOVA was performed on natural logarithm transformed Cmax with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of Cmax for Regimen C (test) versus Regimen D (reference); p = 0.124, ANOVA; LSM difference = 0.9257, 90% CI 2-sided [0.8523 to 1.0053]

2. Primary Outcome: AUC(0-72): Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours Postdose for Alogliptin and Pioglitazone
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK analysis set included all participants in the safety set who had sufficient plasma concentration data to facilitate the derivation of at least 1 PK parameter.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 70 | 69 | 68 | 70
hour*nanogram per milliliter (h*ng/mL)
  Alogliptin | 2197.3 (340.92) | 2163.4 (362.83) | 2194.7 (379.27) | 2195.0 (379.80)
  Pioglitazone | 5726.0 (1826.18) | 5471.9 (1766.76) | 10141.6 (3611.38) | 9907.6 (3495.57)
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; Test type: Equivalence — Alogliptin: For each analyte, ANOVA was performed on natural logarithm transformed AUC(0-72) with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of Cmax for Regimen A (test) versus Regimen B (reference); p = 0.081, ANOVA; LSM difference = 1.0157, 90% CI 2-sided [1.0009 to 1.0308]
Statistical Analysis 2: Comparison: Regimen C vs Regimen D; Test type: Equivalence — Alogliptin: For each analyte, ANOVA was performed on natural logarithm transformed AUC(0-72) with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of AUC(0-72) for Regimen C (test) versus Regimen D (reference); p = 0.922, ANOVA; LSM difference = 1.0009, 90% CI 2-sided [0.9862 to 1.0158]
Statistical Analysis 3: Comparison: Regimen A vs Regimen B; Test type: Equivalence — Pioglitazone: For each analyte, ANOVA was performed on natural logarithm transformed AUC(0-72) with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of AUC(0-72) for Regimen A (test) versus Regimen B (reference); p = 0.066, ANOVA; LSM difference = 1.0486, 90% CI 2-sided [1.0051 to 1.0939]
Statistical Analysis 4: Comparison: Regimen C vs Regimen D; Test type: Equivalence — Pioglitazone: For each analyte, ANOVA was performed on natural logarithm transformed AUC(0-72) with factors for sequence, the participant nested within sequence, period, and regimen. For the relative BA determination, pairwise comparisons were performed to assess the relative BA of alogliptin and pioglitazone via point estimates and 90% CI for the ratio of AUC(0-72) for Regimen C (test) versus Regimen D (reference); p = 0.308, ANOVA; LSM difference = 1.0267, 90% CI 2-sided [0.9839 to 1.0714]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug and no more than 14 days (approximately Day 35) or 30 days (approximately Day 51) for a serious adverse event after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Regimen A | Regimen B | Regimen C | Regimen D
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69 | 0/68 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69 | 0/68 | 0/70
Other Adverse Events (participants affected / at risk) | 2/70 | 1/69 | 1/68 | 2/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (N=70) | Regimen B (N=69) | Regimen C (N=68) | Regimen D (N=70)
Allergic oedema (Immune system disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT03501277/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03501277/SAP_001.pdf